CLINICAL TRIAL: NCT04760210
Title: Compare the Effects of Decompression With ELDOA on Lumbar Disc Protrusion Patient
Brief Title: Decompression With ELDOA on Lumbar Disc Protrusion Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aqua Medical Services (Pvt) Ltd (Industry)
Responsible Party: Principal Investigator, Mir Arif Hussain, Assistant Professor, Aqua Medical Services (Pvt) Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC 00492 Abdul Ghafoor
Record Dates: First submitted 2021-02-04; First posted 2021-02-18 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Lumbar Disc Herniation; Spinal Disk Injury; Protrusion
Keywords: Lumbar Disc Protrusion; Spinal Decompression; Rehabilitation
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Pre-physiotherapy session:
  1. Tens
  2. Infrared/Moist Heat heat for 10 minutes at the low back region.
  3. Lumbar Mobilization (Maitland) CPA 3 sets of 10 reps
  4. Stretching Exercises (Calf, Hams, Back Extensors) 3 sets of 8-10 reps
  5. Strengthening Exercises (Back Extensors) 3 sets of 8-10 reps
  6. Postural Education
  7. Home Plan with lumbar Sacral Support
  Bed rest after the controlled treatment is recommended for this group.
  Interventions: Other: Control Group
- Decompression (Active Comparator): Pre-physiotherapy session:
  1. Tens
  2. Infrared/Moist Heat heat for 10 minutes at the low back region.
  3. Lumbar Mobilization (Maitland) CPA 3 sets of 10 reps
  4. Stretching Exercises (Calf, Hams, Back Extensors) 3 sets of 8-10 reps
  5. Strengthening Exercises (Back Extensors) 3 sets of 8-10 reps
  6. Postural Education
  7. Home Plan
  Decompression therapy session after the controlled treatment is recommended for this group.
  Interventions: Other: Decompression Group
- ELDOA (Active Comparator): Pre-physiotherapy session:
  1. Tens
  2. Infrared/Moist Heat heat for 10 minutes at low back region.
  3. Lumbar Mobilization (Maitland) CPA 3 sets of 10 reps
  4. Stretching Exercises (Calf, Hams, Back Extensors) 3 sets of 8-10 reps
  5. Strengthening Exercises (Back Extensors) 3 sets of 8-10 reps
  6. Postural Education
  7. Home Plan
  Segmental Spinal ELDOA Exercise after the controlled treatment is recommended for this group.
  Interventions: Other: ELDOA

INTERVENTIONS:
Other: Control Group — Treatment for this group is conventional physical therapy along with the bed rest.
  Other Names: Group A
  Arms: Control Group
Other: Decompression Group — Treatment for this is conventional physical therapy along with the spinal decompression.
  Other Names: Group B
  Arms: Decompression
Other: ELDOA — Treatment for this is conventional physical therapy along with the ELDOA.
  Other Names: Group C
  Arms: ELDOA

SUMMARY:
Decompression therapy is a result-oriented approach but it expensive and minimum availability in Pakistan. In physical therapy, we use different exercises to solve multiple spine problems. Some exercises used to treat orthogenic components such as mobilization, manipulation, SNAGS, and traction. Some exercises used to treat myogenic components such as muscle energy technique, neuromuscular reeducation, active isolated stretch, etc. Some exercises used to treat neurogenic components such as Neurodynamics, Active release technique, etc. As we know the fascia is an important component in our body most of the time the fascia restriction makes the patient condition verse. A researcher introduced the systems of exercise more the 35 years ago which works especially on the spine at every intervertebral level including costal and pelvic articulation. These exercises are called Elongation Longitudinaux Avec Decoaption Osteo-Articulaire (ELDOA) or simply Longitudinal Osteo-Articular De-coaptation Stretching (LOADS). It can be described as a fascial stretch that's localized tension at the level of a specific spinal segment and create decompression. In which he combined improving the tone of the intrinsic muscles of the spine along with reinforcing the extrinsic muscles related to the spine aim the back and stretching the interlinking paraspinal muscles. ELDOA exercise is designed for every level of the spine from the base of the skull to the sacroiliac joint. In each ELDOA exercise, we create fascial tension above and below the joint or disc that one is trying to "open up" or decompress. The outcomes include; Release vertebral compression, improved blood circulation, Disc re-hydration, improve muscle tone, and awareness. One of my studies also proved that ELDOA Exercises improve the pain and functional level in spinal disc protrusion patients.

DETAILED DESCRIPTION:
Low back pain is the common problem of our society, 80% of people experience back pain at some stage of their life. Low Back pain lifetime prevalence is 65% to 80% and It is estimated that 28% experience disabling low back pain sometime during their lives. Point prevalence ranged from 12% to 33%, the 1-year prevalence ranged from 22% to 65%, and lifetime prevalence ranged from 11% to 84%. Back pain peak prevalence age is 40-50, First episode of start in the '20s and recurrence rates between 39-71%. Women tend to be affected more in cervical spine problems than men and men tend to more affected in lumbar spine problems than women. The majority (80-90%) of low back disorders occur at the L4/5 and/or L5/S1. The occupational risk factor include driving (P<0.001), lifting, carrying, pulling, pushing, and twisting (P<0.001 for all variables) as well as nondriving vibrational exposure (P<0.001).

Maitland divides lumbar spine problems into two groups, in the first group the L4/5 and L5/S1 intervertebral discs are frequently a source of symptoms and the second group has postural, muscle balance, muscle weakness, muscles spasm degenerative changes, and mechanical movement disorders problems. The L5-S1 Segment is the most common site of problem in the spine because this level bears more weight, Center of gravity passes directly through this vertebra, transition L5 Mobile and S1 Stable, Large angle B/w L5 & S1 and a great amount of movement.

The intervertebral disk makes up 1/3 of the total length of the vertebral column. The disc contains 85% to 90% of water, but the amount decreases up to 65% with age. The water-binding capacity of the disc decrease with age and degenerative changes begin to occur after 2nd decade of life. The Facet joint carries 20-25% axial body load but this may reach 70% with degeneration of the Disc. The most significant biochemical change to occur in disc degeneration is the loss of proteoglycan. This loss is responsible for a fall in the osmotic pressure of the disc matrix and therefore a loss of hydration. Loading may thus lead to inappropriate stress concentrations along the endplate or in the annulus.

CT Classification of Annular Tears There are five possible severities of the radial annular tear as seen on an axial CT image.

* The grade 0 is a normal disc, where no contrast material injected in the center of the disc has leaked from the confines of the nucleus pulposus.
* The grade 1 tear has leaked contrast material but only into the inner one-third of the annulus.
* In the grade 2 tear, the contrast has leaked from the nucleus into the outer two-thirds of the annulus.
* The grade 3 tear has leaked contrast completely through all three zones of the annulus.
* The grade 4 tear the contrast has spread circumferentially around the disc, often resembling a ship's anchor. Pathologically, this represents the merging of a full-thickness radial tear with a concentric annular tear.
* The grade 5 tear completely ruptured the outer layers of the disc and is leaking contrast material from the disc into the epidural space. This type of tear is thought to have the ability to induce a severe inflammatory reaction in the adjacent neural structures. In some patients, this inflammatory process is so severe that it causes painful chemical radiculopathy and sciatica without the presence of nerve root compression.

Low-back pain with leg pain may be caused by a herniated intervertebral disc exerting pressure on the nerve root. Most patients will respond to conservative treatment, but in carefully selected patients, a surgical discectomy may provide faster relief of symptoms. The Patient's history and physical examination along with MRI confirm the disc herniation diagnosis. In the case of spinal disc herniation, the management is Surgical and conservative. In surgery, we have percutaneous procedures such as chymopapain injections, Annuloplasty, Percutaneous disc decompression, and Endoscopic percutaneous discectomy and Open Surgery such as Laminectomy, Discectomy/Microdiscectomy, Artificial disc surgery, and Spinal fusion. The Conservative Management includes Oral Analgesic, Gentle traction, Spinal Decompression, Spinal Stabilization, Exercise, and Fascia Stretching (ELDOA).

ELIGIBILITY:
Inclusion Criteria:

* MRI of the lumbar spine showing lumbar disc bulge
* Localized and radiating pain more than 5 on NPRS

Exclusion Criteria:

* Lumbar spondylolisthesis
* Spinal stenosis
* Fracture of the lumbar spine
* Spinal tumor
* Ankylosing spondylitis
* Patients taking blood thinner medication

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Up to 3 weeks
  The scale of pain. The patient will be asked to report pain on a 1-10 numbering scale. 1 means minimum pain and 10 means extreme pain.
Oswestry disability index | Up to 3 weeks
  The scale of disability. The patient will be asked the referenced questions and the assessor will tick the answers. The maximum score of the Oswestry disability index is 100 percent which means complete disability whereas the minimum score is 0 percent which means no disability at all.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ghafoor Sajjad, MSPT, Principal Investigator — Shifa Tameer-e-Millat University Islamabad
Locations (1):
- Aqua research Center, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Archaeos Projects. (1999). Preliminary Site Report of the Oriental Institute of the University of Vienna and Archaeos: Excavation Project at Tell Arbid, Sector D Retrieved 04/09/2004, 2004, from http://www.archaeos.org/html/repor2js.htm
- [Background] Atlas SJ, Keller RB, Wu YA, Deyo RA, Singer DE. Long-term outcomes of surgical and nonsurgical management of lumbar spinal stenosis: 8 to 10 year results from the maine lumbar spine study. Spine (Phila Pa 1976). 2005 Apr 15;30(8):936-43. doi: 10.1097/01.brs.0000158953.57966.c0. PMID 15834339
- [Background] Breslau, A. M., & Gabe, M. (1962). Ergebnisse der Polysaccharidhistochemie, Microorganismen, Invertebraten : mit 25. Stuttgart: Fischer.
- [Background] Delauche-Cavallier MC, Budet C, Laredo JD, Debie B, Wybier M, Dorfmann H, Ballner I. Lumbar disc herniation. Computed tomography scan changes after conservative treatment of nerve root compression. Spine (Phila Pa 1976). 1992 Aug;17(8):927-33. PMID 1387974
- [Background] Dvorak J, Gauchat MH, Valach L. The outcome of surgery for lumbar disc herniation. I. A 4-17 years' follow-up with emphasis on somatic aspects. Spine (Phila Pa 1976). 1988 Dec;13(12):1418-22. doi: 10.1097/00007632-198812000-00015. PMID 3212575
- [Background] Frymoyer JW, Pope MH, Costanza MC, Rosen JC, Goggin JE, Wilder DG. Epidemiologic studies of low-back pain. Spine (Phila Pa 1976). 1980 Sep-Oct;5(5):419-23. doi: 10.1097/00007632-198009000-00005. PMID 6450452
- [Background] Hammer, W. I. (2007). Functional soft-tissue examination and treatment by manual methods: Jones & Bartlett Learning.
- [Background] Khan, A. G. S. G. A., & Khan, A. (2016). Fascia Stretching Improve the Pain and Functional Level in Disc Protrusion Patients. Journal of Riphah College of Rehabilitaion Sciences, 4(1), 7-10.
- [Background] Krause M, Refshauge KM, Dessen M, Boland R. Lumbar spine traction: evaluation of effects and recommended application for treatment. Man Ther. 2000 May;5(2):72-81. doi: 10.1054/math.2000.0235. PMID 10903582
- [Background] Saal JA, Saal JS. Nonoperative treatment of herniated lumbar intervertebral disc with radiculopathy. An outcome study. Spine (Phila Pa 1976). 1989 Apr;14(4):431-7. doi: 10.1097/00007632-198904000-00018. PMID 2718047
- [Background] van der Windt DA, Simons E, Riphagen II, Ammendolia C, Verhagen AP, Laslett M, Deville W, Deyo RA, Bouter LM, de Vet HC, Aertgeerts B. Physical examination for lumbar radiculopathy due to disc herniation in patients with low-back pain. Cochrane Database Syst Rev. 2010 Feb 17;(2):CD007431. doi: 10.1002/14651858.CD007431.pub2. PMID 20166095
- [Background] Weber H. Lumbar disc herniation. A controlled, prospective study with ten years of observation. Spine (Phila Pa 1976). 1983 Mar;8(2):131-40. PMID 6857385